CLINICAL TRIAL: NCT01939925
Title: Communicating Evidence From Systematic Reviews to the Public: A Randomised Controlled Trial
Brief Title: Communicating Evidence From Systematic Reviews to the Public
Acronym: PLSRCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian Knowledge Centre for the Health Services (Other Government)
Collaborators: McMaster University (Other); University of Ottawa (Other); Asociacion Colaboracion Cochrane Iberoamericana (Other); University of Milan (Other)
Responsible Party: Principal Investigator, Claire Glenton, Senior Researcher, Norwegian Knowledge Centre for the Health Services
Allocation: Randomized | Model: Parallel | Masking: Quadruple
Other Study IDs: PLSRCT1
Record Dates: First submitted 2013-08-27; First posted 2013-09-11 (Estimated); Last update posted 2013-09-11 (Estimated); Status verified 2013-09

CONDITIONS: Adult
Keywords: patient education; Health Knowledge, Attitudes, Practice; comprehension; consumer health information
MeSH Terms: conditions — Behavior

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- New plain language summary format (Experimental): New plain language summary format of a Cochrane systematic review
  Interventions: Other: New plain language summary format
- Current plain language summary format (Active Comparator): Plain Language Summary format for the public currently in use in Cochrane systematic reviews
  Interventions: Other: Current plain language summary format

INTERVENTIONS:
Other: New plain language summary format — New plain language summary includes qualitative and quantitative description of text (absolute effects and natural frequencies provided); quantitative results provided in a table; quality of the evidence according to GRADE provided in a table; question and answer format; follows principles of linguistic frameworks (e.g. progressive movements from introduction to 'bottom line')
  Arms: New plain language summary format
Other: Current plain language summary format — Current plain language summary includes qualitative description of effects only; inconsistent description of the quality of the evidence; paragraph of text; inconsistent flow of information
  Arms: Current plain language summary format

SUMMARY:
The purpose of this randomised controlled trial is to compare a new standardised summary format for presentation of synthesised evidence from systematic reviews for the public (a new plain language summary format) to the current format used in Cochrane systematic reviews. The study will evaluate if the new presentation improves understanding about the benefits and harms of an intervention, if it improves the accessibility of the information, and if it is preferred over other versions by the public over the current format.

ELIGIBILITY:
Inclusion Criteria:

* patients or members of the public 16 years or older

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 193 (Actual)
Dates: Start 2009-05; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Understanding of benefits and harms | After reading summary - time 0
  Average proportion of people who answered 5 multiple choice questions correctly. Each question includes five response options about the number of people who could benefit or be harmed by the intervention and about the quality of evidence

SECONDARY OUTCOMES:
Number of questions answered correctly | After reading summary - time 0
  Total number of questions out of five questions for benefits and harms that were answered correctly

OTHER OUTCOMES:
Understanding of the purpose of the summary | after reading summary - time 0
  A multiple choice question with three options
Understanding the producer of the summary | after reading summary - time 0
  A multiple choice question with three options
Usability and accessibility | after reading summary - time 0
  Five questions about whether information was easy to find and understand, reliable, and useful to someone making a decision. Measured using a 7 point Likert scale (strongly agree to strongly disagree).
Preference for the new format or the old format | after reading both summaries - time 0
  7 point likert scale

CONTACTS AND LOCATIONS:
Overall Officials: Claire Glenton, PhD, Principal Investigator — Norwegian Knowledge Centre for the Health Services; Holger J Schunemann, MD PhD, Principal Investigator — McMaster University; Nancy A Santesso, RD PhD cand, Principal Investigator — McMaster University
Locations (5):
- Argentine Cochrane Centre, Instituto de Efectividad Clínica y Sanitaria (IECS), Buenos Aires, Argentina
- University of Ottawa, Ottawa, Ontario, Canada
- University of Milan, Milan, Italy
- Norwegian Knowledge Centre for the Health Services, Oslo, Norway
- Centro Cochrane Iberoamericano - Hospital de la Santa Creu i Sant Pau, Barcelona, Spain